CLINICAL TRIAL: NCT03871790
Title: Peptide-based Immunization for Colon- and Pancreas-carcinoma (PICOP-GLOBAL): An International, Multicenter Protocol
Brief Title: Peptide-based Immunization for Colon- and and Pancreas-carcinoma
Acronym: PICOP-GLOBAL
Status: Completed | Type: Observational
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: PICOP-GLOBAL-2019
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Colon Neoplasm; Colon Adenocarcinoma; Colon Cancer; Colo-rectal Cancer; Rectal Cancer; Rectal Neoplasms; Rectal Adenocarcinoma; Rectal Tumors; Pancreatic Cancer; Pancreas Cancer; Pancreatic Neoplasms; Pancreatic Adenocarcinoma
Keywords: Neoepitopes; Vaccination; Tumor-specific antigens; Personalized medicine
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood in EDTA tube, blood in Cell-free DNA tube (Streck tube), and blood in Heparin tube
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with colorectal cancer: Participants with colorectal cancer ongoing surgery older than 18 years old.
- Participants with pancreatic cancer: Participants with pancreatic cancer ongoing surgery older than 18 years old.

SUMMARY:
An international, multicenter study to identify tumor molecular particularities and neoepitopes among participants with colorectal and pancreatic tumors undergoing surgery.

DETAILED DESCRIPTION:
Colorectal and pancreatic cancers are among the most common causes of cancer-related death over the world. Standard of care treatment for colon and pancreas cancer is stage dependent and includes surgical, chemotherapeutic, and radiation therapy. However, the current statistics underlines an urgent need for improved treatment. Patient-individualized treatments and enhancement of the immune response via vaccination are among new therapeutic options.

The enhancement of the immune response via vaccination is among new therapeutic options. Here, either cell-specific antigens, over-expressed tumor specific antigens or mutated tumor-specific antigens (neoepitopes) can be employed. Especially the latter possess the biggest potential for high specificity but presuppose an extensive characterization of the respective tumor. In order to identify a neoepitope-based vaccination approach for patient-individualized treatment options the molecular particularities of tumors have to be analysed.

The aim of this study is to identify tumor molecular particularities and neoepitopes among patients with colorectal and pancreatic tumors undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent is obtained from the participant
* Patients with pancreas or colorectal carcinoma undergoing surgery
* The participant is older than 18 years old

Exclusion Criteria:

* Inability to provide informed consent
* The patient is not suffering from pancreas or colo-rectal carcinoma
* Patient has a condition contradicting surgery
* The participant is younger than 18 years old
* Previously enrolled in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal or pancreas carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Identification of tumor specific mutations on the genomic level | 24 months
  Identification of tumor specific mutations on the genomic level using whole exome sequencing and/or whole genome sequencing

SECONDARY OUTCOMES:
Identification of tumor specific mutations on transcriptional and/or translational level | 24 months
  Direct comparison of tumor and non-tumor tissue to identify somatic mutations through RNA sequencing and proteomics analysis
Identification of neo-antigens epitopes at protein level | 24 months
  Identification of neo-antigens epitopes at protein level via mass spectrography

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Principal Investigator — CENTOGENE GmbH Rostock
Locations (1):
- Teaching Hospital UOL Cancer Center, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bobisse S, Genolet R, Roberti A, Tanyi JL, Racle J, Stevenson BJ, Iseli C, Michel A, Le Bitoux MA, Guillaume P, Schmidt J, Bianchi V, Dangaj D, Fenwick C, Derre L, Xenarios I, Michielin O, Romero P, Monos DS, Zoete V, Gfeller D, Kandalaft LE, Coukos G, Harari A. Sensitive and frequent identification of high avidity neo-epitope specific CD8 + T cells in immunotherapy-naive ovarian cancer. Nat Commun. 2018 Mar 15;9(1):1092. doi: 10.1038/s41467-018-03301-0. PMID 29545564
- [Background] Bousquet G, Janin A. Patient-Derived Xenograft: An Adjuvant Technology for the Treatment of Metastatic Disease. Pathobiology. 2016;83(4):170-6. doi: 10.1159/000444533. Epub 2016 Mar 25. PMID 27010922
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Cho YT, Su H, Wu WJ, Wu DC, Hou MF, Kuo CH, Shiea J. Biomarker Characterization by MALDI-TOF/MS. Adv Clin Chem. 2015;69:209-54. doi: 10.1016/bs.acc.2015.01.001. Epub 2015 Feb 17. PMID 25934363
- [Background] Dangles-Marie V, Pocard M, Richon S, Weiswald LB, Assayag F, Saulnier P, Judde JG, Janneau JL, Auger N, Validire P, Dutrillaux B, Praz F, Bellet D, Poupon MF. Establishment of human colon cancer cell lines from fresh tumors versus xenografts: comparison of success rate and cell line features. Cancer Res. 2007 Jan 1;67(1):398-407. doi: 10.1158/0008-5472.CAN-06-0594. PMID 17210723
- [Background] Maule M, Merletti F. Cancer transition and priorities for cancer control. Lancet Oncol. 2012 Aug;13(8):745-6. doi: 10.1016/S1470-2045(12)70268-1. No abstract available. PMID 22846827
- [Background] Murtaza M, Dawson SJ, Tsui DW, Gale D, Forshew T, Piskorz AM, Parkinson C, Chin SF, Kingsbury Z, Wong AS, Marass F, Humphray S, Hadfield J, Bentley D, Chin TM, Brenton JD, Caldas C, Rosenfeld N. Non-invasive analysis of acquired resistance to cancer therapy by sequencing of plasma DNA. Nature. 2013 May 2;497(7447):108-12. doi: 10.1038/nature12065. Epub 2013 Apr 7. PMID 23563269
- [Background] Philip PA, Mooney M, Jaffe D, Eckhardt G, Moore M, Meropol N, Emens L, O'Reilly E, Korc M, Ellis L, Benedetti J, Rothenberg M, Willett C, Tempero M, Lowy A, Abbruzzese J, Simeone D, Hingorani S, Berlin J, Tepper J. Consensus report of the national cancer institute clinical trials planning meeting on pancreas cancer treatment. J Clin Oncol. 2009 Nov 20;27(33):5660-9. doi: 10.1200/JCO.2009.21.9022. Epub 2009 Oct 26. PMID 19858397
- [Background] Pompili L, Porru M, Caruso C, Biroccio A, Leonetti C. Patient-derived xenografts: a relevant preclinical model for drug development. J Exp Clin Cancer Res. 2016 Dec 5;35(1):189. doi: 10.1186/s13046-016-0462-4. PMID 27919280
- [Background] Rammensee HG, Singh-Jasuja H. HLA ligandome tumor antigen discovery for personalized vaccine approach. Expert Rev Vaccines. 2013 Oct;12(10):1211-7. doi: 10.1586/14760584.2013.836911. Epub 2013 Oct 4. PMID 24090147
- [Background] Shaw JA, Stebbing J. Circulating free DNA in the management of breast cancer. Ann Transl Med. 2014 Jan;2(1):3. doi: 10.3978/j.issn.2305-5839.2013.06.06. PMID 25332979